CLINICAL TRIAL: NCT02502695
Title: A Prospective, Observational, Quality Improvement Study to Optimize Care for Lung Cancer Patients Undergoing Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: A Study to Optimize Care for Lung Cancer Patients Undergoing Video-Assisted Thoracoscopic Surgery (VATS)
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Scott J. Swanson, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 15-193
Record Dates: First submitted 2015-06-26; First posted 2015-07-20 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
Keywords: VATS Lobectomy and Segmentectomy for Lung Cancer; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1-VATS-associated best practices: * Data to be collected will include demographic data and information about the pre-operative workup, surgical procedure, postoperative course and early discharge course for these patients.
  * After the last patient completes the 30-day post surgery follow-up, the investigators will determine a set of best practices to implement at each of the sites for the quality improvement initiative. During the assessment period, no patients will be enrolled into the study.
  Interventions: Other: VATS-associated best practices
- Cohort 2-VATS-associated best practices: -Once the set of VATS-associated best practices, an additional cohort of approximately 200 patients will be enrolled and followed in a manner identical to the first cohort.
  Interventions: Other: VATS-associated best practices

INTERVENTIONS:
Other: VATS-associated best practices

SUMMARY:
This is a research study for participants who have been diagnosed with lung cancer and are receiving VATS (Video Assisted Thoracoscopic Surgery) lobectomy or segmentectomy. The overall objective of this study is to develop a database to collect data on participants who are undergoing VATS lobectomy or segmentectomy for lung cancer.

DETAILED DESCRIPTION:
This database will be used as for quality improvement purposes. Furthermore, the database will help in collecting data in an organized fashion, which will help the investigators learn more about the details of the workup performed prior to the surgery, during the surgery, peri-operative management and early follow-up. The investigators hope that this database will help to determine a common guideline to perform VATS lobectomy or segmentectomy. By creating a common guideline for future treatment of VATS patients, the investigators predict the efficiency of the process will increase significantly without decreasing, and perhaps even improving, the quality of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age ≥ 18 years
* Underwent a VATS lobectomy or segmentectomy procedure for lung cancer -- Note: patients with other malignancies are eligible if they have a primary cancer of the lung as defined above

Exclusion Criteria:

* Subjects undergoing thoracotomy lobectomy or segmentectomy for lung cancer
* Subjects undergoing surgical procedures other than VATS lobectomy or segmentectomy for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that will have VATS lobectomy and segmentectomy procedures for lung cancer
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Readmissions rates within 30 days of the patient's surgery date | 30 Days
Incidence of post-operative complications within 30 days of the patient's surgery date | 30 Days
Total inpatient cost | 30 Days

SECONDARY OUTCOMES:
Difference in readmission rates between the two cohorts | 3 years
  To compare current VATS-associated procedures with a set of best VATS-associated practives implemented across the participating study centers

CONTACTS AND LOCATIONS:
Overall Officials: Scott J. Swanson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (6):
- United States (6):
  - Providence Saint John's Health Center, Santa Monica, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - WellStar Medical Group, Austell, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri